CLINICAL TRIAL: NCT01976910
Title: A Protocol for the Safety and Tolerance of Intravenous 4-Demethylcholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) in Patients With Advanced Cancer
Brief Title: Study of 4-Demethylcholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) in Patients With Advanced Cancer"
Acronym: DM-CHOC-PEN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DEKK-TEC, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68,876; 5R43CA132257-02 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-06 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Advanced Cancer
Keywords: Advanced cancers; Brain Neoplasms, Malignant, Primary; Brain Tumor, Recurrent; Advanced cancer
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 4-DM-CHOC-PEN (Experimental): DM-CHOC-PEN is an intervention and will be dosed @ 39 mg/M2,escalated in 1-patient cohorts at 40% dosage.
  * At the 1st DLT - expand to 3-6 patient cohorts/dose with escalations at 33% increments.
  * The MTD will be where 2 DLTs are noted and the study is discontinued.
  Interventions: Drug: DM-CHOC-PEN

INTERVENTIONS:
Drug: DM-CHOC-PEN — DM-CHOC-PEN will be dosed @ 39 mg/M2, escalated in 1-patient cohorts at 40% dosage.
  At the 1st DLT - expand to 3-6 patient cohorts/dose with escalations at 33% increments.
  The MTD will be where 2 DLTs are noted and the study is discontinued.
  Other Names: 4-Demethylcholesteryloxycarbonylpenclomedine

SUMMARY:
DM-CHOC-PEN is a polychlorinated pyridine cholesteryl carbonate that has demonstrated antineoplastic activities in human xenograft intracerebrally implanted tumor mouse models, acceptable preclinical toxicities in mouse, rat and dog models; and no behavioral cognitive impairment/neurotoxicities were noted in mouse and rat models.

The drug is ready for human use as an soy bean oil/lecithin/glycerin water emulsion, the latter which has been documented - chemically and biologically to be stable and safe. Patients are currently being enrolled and treated with the protocol.

Patients with advanced cancer, with or without central nervous system involvement will be eligible for enrollment, providing the required blood and other eligibility requirements are met.

DETAILED DESCRIPTION:
4-Demethylcholesterylpenclomedine(DM-CHOC-PEN)is a polychlorinated pyridine cholesteryl carbonate that has demonstrated complete remissions when administrated to mice bearing intracranially implanted human cancer xenografts (glioblastomas and breast cancers) and has acceptable preclinical toxicity profiles - mice, rats and dogs.

The drug is being administered intravenously once every 21 days as an infusion. The starting dose was 39 mg/M2 (based on 1/10 LD10 observed in mice and rats).

A modified accelerated dosing protocol of Simon, Freidlin, et al is in process to escalate dosage which will reduce the number of patients required and minimize ineffective doses. The protocol will result in one patient cohorts at 40% dosage escalations. When the 1st instance of a dose limiting toxicity (DLT) [grade - 3 or 4 toxicity] is observed, or the 2nd instance of a 1st course grade 2 toxicity of any type is observed, the cohort for that current dose level will be expanded to 3-6 patients and escalation will proceed at 33% increments.

During the entirety of the study, intra-patient escalation will be allowed. This will occur if the patient experiences are < grade 2 toxicity at the existing dose, if no > grade 2 toxicity was identified at the existing dose and no DLTs were noted at the higher dose level (if any patients had been escalated to that dose).

Continuation of therapy - Patients who experience stabilization, partial or complete remission while being treated will continue to receive the drug as per the last dose prior to identifying positive results at an every 3 weeks interval.

Discontinuation of therapy - progressive disease and/or toxicities.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histological evidence of a solid malignant tumor (hematological malignancies are excluded) with convincing clinical, radiographic or isotopic evidence of cancer, for which no effective proven treatment exists. CNS associated tumors are preferred, but not required. Patients must sign an informed consent that complies with the investigator/DEKK-TEC policies and approved by a Human Investigation Review Committee.
* All patients must have a projected survival time of at least 12 weeks and a Karnofsky performance score: >60% (or Zubrod score of >2).
* All patients must be off previous chemo- and/or radiotherapy for at least three (3) weeks prior to entrance into the study and have recovered from any toxic effects induced by such treatment(s). Patients who have received a nitrosourea type drug must have had no treatment within the last six weeks.
* Measurable lesions are not required for admittance to the study - but are desirable.
* Age initiated after limitation - 18 years or older. A separate pediatric study is proposed to evaluate tolerance to the drug in children.
* Gender is not a criterion.

Exclusion Criteria:

* Hematology WBC <4,000 mm3 Platelets <100,000 mm3
* Liver Function If bilirubin, AST, and/or ALT are >ULN
* Renal Function Creatinine >1.5 mg%
* Cardiovascular Acute myocardial infarction Congestive heart failure - (NYHA criteria for uncontrolled) Clinically significant cardiac arrhythmias - uncontrolled
* Concomitant chemotherapy or radiotherapy is not permitted.
* Pregnant or lactating females are excluded. Women of childbearing age, and their sexual partners, must use an effective contraception program. Males who are having sexual relations with women capable of child bearing must use birth control while on the study and for 3-months after the last dose of the study drug.
* Allergies to eggs, lecithin or soy products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hyperbilirubinemia | 3-year
  Document hepatic toxicity.

SECONDARY OUTCOMES:
Document a MTD | 2-3 years
  Patients were treated in cohorts from 39-111 mg/m2 single IV doses. Hepatic toxicity was a limiting factor for patients w/ liver disease.
  Phase II trials will be 2-tier - w/ liver involvement and without,.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus L Ware, MD, Principal Investigator — Tulane University Medical School
Locations (1):
- Tulane University Medical School, New Orleans, Louisiana, United States

REFERENCES:
- See also: Related Info — http://dekk-tec.com